CLINICAL TRIAL: NCT06667115
Title: The Effectiveness of Proprioceptive Neuromuscular Facilitation Exercise With Virtual Reality Motion Capture Gaming System and Concurrent Feedback on Early Shoulder Muscle Activation in Healthy Individuals
Brief Title: Proprioceptive Neuromuscular Facilitation Exercise on Early Shoulder Muscle Activation in Healthy Individuals
Acronym: PNF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dominican University New York (Other)
Responsible Party: Principal Investigator, Ayse Edeer, Principal investigator, Dominican University New York
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Dominican University New York
Record Dates: First submitted 2024-10-28; First posted 2024-10-31 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Exercise; Healthy
Keywords: proprioceptive neuromuscular facilitation; virtual reality; concurrent feedback; shoulder; muscle activation
MeSH Terms: conditions — Motor Activity | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF and PNF with virtual reality and PNF with concurrent feedback (Active Comparator): Participants began with the PNF D2 shoulder exercise for 1 minute. Then participants did PNF D2 exercise with virtual reality gaming as second intervention for 1 minute and then they did PNF D2 exercise with concurrent feedback as third intervention for 1 minute. Between each intervention, participants were given a 2-minute break. Baseline was always PNF exercise, however second and third interventions for the arm 1 and arm 2 were different.
  Interventions: Other: PNF exercise; Other: PNF exercise with virtual reality gaming; Other: PNF with concurrent feedback
- PNF and PNF with concurrent feedback and PNF with virtual reality gaming (Active Comparator): Participants began with the PNF D2 shoulder exercise for 1 minute. Then participants did PNF D2 exercise with concurrent feedback as second intervention for 1 minute and then they did PNF D2 exercise with virtual reality gaming as third intervention for 1 minute. Between each intervention, participants were given a 2-minute break. Baseline was always PNF exercise, however second and third interventions for the arm 1 and arm 2 were different.
  Interventions: Other: PNF exercise; Other: PNF exercise with virtual reality gaming; Other: PNF with concurrent feedback

INTERVENTIONS:
Other: PNF exercise — Foundational PNF D2 shoulder flexion exercise incorporating shoulder flexion, abduction, and external rotation. This exercise was performed at a metronome-guided pace of 14 beats per minute to establish a consistent baseline.
Other: PNF exercise with virtual reality gaming — Combined the PNF D2 shoulder flexion exercise with a virtual reality motion capture game (the U-Ball game).
Other: PNF with concurrent feedback — PNF exercise with the addition of auditory concurrent feedback ("Sword") which referenced the action of unsheathing a sword in a diagonal upward direction.

SUMMARY:
The study explores the effect of proprioceptive neuromuscular facilitation (PNF) exercises combined with virtual reality (VR) motion capture system and concurrent feedback (CF), on early shoulder muscle activation in healthy individuals. Thirty healthy individuals performed three PNF D2 shoulder exercises sequentially: first PNF alone, then PNF with VR (using U-Ball game (BeCure Global Inc.) on Xbox Kinect (PNF+VR), and PNF with VR and CF (PNF+VR+CF), with the latter two in a randomized order. Using wireless surface electromyography (EMG) and 3D inertial measurement units (Noraxon USA, Inc.), the activation of the upper trapezius (UT), lower trapezius (LT), infraspinatus (INF), and serratus anterior muscles (SA), along with shoulder flexion, abduction, and external rotation range of motion were recorded during three shoulder exercises.

DETAILED DESCRIPTION:
Study Design A one-way repeated measures design was employed to investigate the potential benefits of augmenting PNF exercises with VR and concurrent feedback for enhancing early shoulder muscle activation in healthy individuals.

Participants Thirty healthy volunteers (14 males and 16 females with an average age of 26.2 ± 4 years) were recruited through convenience sampling. The inclusion criteria required being 18-45 years old and capable of performing PNF D2 shoulder flexion exercise. Exclusion criteria, designed to ensure sample homogeneity and data reliability, included any shoulder injuries in the dominant arm within the last 3 months, such as pain in the scapular region, rotator cuff tear or reconstruction, shoulder dislocation, shoulder instability, frozen shoulder, fracture, and chronic neck pain. This study received ethical approval from the Institutional Review Board (IRB) as minimal risk research (IRB # 2023-0322-01). The study protocol conforms to the ethical guidelines of the 1975 Declaration of Helsinki (Helsinki Declaration as revised in 2013).

Researchers screened potential participants for inclusion criteria. Eligible individuals were given a detailed explanation of the study's purpose, interventions, and their role, followed by informed consent. Participants then completed a demographic information form. To protect confidentiality, participants were assigned numerical identifiers, and all identifying information was stored separately from research data in a secure location.

Outcome measures This study utilized a combination of technologies to measure shoulder muscle activation and ROM. The NORAXON 3D Motion Capture system, equipped with Ultium EMG sensors and Ultium Motion sensors, provided precise tracking of muscle activity and movement patterns (ICC ranging from 0.87-0.98). The Ultium surface EMG Sensors were utilized to detect the Maximum Voluntary Contraction (MVC) as well as muscle activation in the form of % MVC during three different interventions. Ultium Motion ROM sensors were utilized to analyze the PNF D2 shoulder flexion exercise in three different planes of motion via flexion, abduction, and external rotation. Data collection was conducted using MyoMUSCLE and MyoMOTION software.

Participants' subjective feedback was collected using the Borg Rating of Perceived Exertion (RPE) scale and a customized questionnaire including enjoyment, confidence, frustration, boredom, and level of difficulty.

Interventions The Xbox Kinect and BeCure game software were utilized for VR exercises. The U-Ball game challenged participants to hit balls coming from random targets on a screen using the PNF D2 shoulder flexion on their dominant arm. The game setting ensured 14 balls appeared within the intervention period. Visual feedback was provided through an on-screen avatar mirroring the participant's movements. While the game displayed score elements, these were excluded from the study analysis to focus on proper exercise form.

This study implemented three distinct shoulder muscle activation interventions. Intervention I (PNF alone): Foundational PNF D2 shoulder flexion exercise, incorporating shoulder flexion, abduction, and external rotation. This exercise was performed at a metronome-guided pace of 14 beats per minute to establish a consistent baseline and match the U-Ball game's tempo. Intervention II (PNF+VR): Combined the PNF D2 shoulder flexion exercise with a VR motion capture game (the U-Ball game). Intervention III (PNF+VR+CF): PNF D2 shoulder flexion exercise combined with the U-Ball game and the addition of auditory concurrent feedback ("Sword") which referenced the action of unsheathing a sword in a diagonal upward direction. Each intervention lasted 60 seconds, followed by a two-minute rest period which included the survey completion.

Procedures EMG and ROM Sensor Placement Surface EMG electrodes were placed on the identified motor points of the upper trapezius (UT), lower trapezius (LT), infraspinatus (INF), and serratus anterior (SA) muscles. ROM sensors were attached to the upper spine (C7/T1), lower spine (T12/L1), and deltoid tuberosity on the participants' dominant arm. Anatomical landmarks utilized for sensor placement were confirmed by the same two researchers for consistency. A male and female researcher assisted with sensor placement to ensure a respectful and comfortable environment.

Introduction to PNF D2 Flexion Exercise At a learning station, participants were introduced to the PNF D2 shoulder flexion exercise and auditory concurrent feedback via a pre-recorded instructional video. In the video the researcher explained how the auditory "Sword" concurrent feedback was utilized. Another researcher then provided a live demonstration, allowing participants to practice the pattern and confirm their understanding.

MVC Measurements and Calibration Researchers conducted MVC tests for baseline muscle activity. Participants exerted maximum effort against manual resistance applied by the researcher who trained to apply consistent resistance across sessions. ROM sensor calibration took place 1.5 meters from the Xbox Kinect camera, aligning participants with the U-Ball game's software requirements for optimal interaction. Subsequently, muscle activation from UT, LT, SA and INF muscles and shoulder ROM (flexion, abduction, and external rotation) were monitored and recorded for one minute using the MyoMUSCLE and MyoMOTION software (Noraxon Inc.) during the three exercises.

Intervention Administration Participants began with the PNF D2 shoulder exercise at 14 beats per minute paced by a metronome to match the tempo of the U-Ball game for 1 minute. After this initial intervention, participants were given a 2-minute break where they completed a survey (Borg and customized questionnaire). Participants were then randomized for interventions II and III. This randomization involved blindly selecting one of two papers marked II or III, designed to minimize carryover effects.

ELIGIBILITY:
Inclusion Criteria:

* being 18-45 years old
* capable of performing PNF D2 shoulder flexion exercise

Exclusion Criteria:

* any shoulder injuries in the dominant arm within the last 3 months
* pain in the scapular region
* rotator cuff tear or reconstruction
* shoulder dislocation
* shoulder instability
* frozen shoulder
* fracture
* chronic neck pain

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
muscle activation | Through study completion, an average of 6 months
  Using wireless surface electromyography (EMG) (Noraxon USA, Inc.), the activation of the upper trapezius (UT), lower trapezius (LT), infraspinatus (INF), and serratus anterior muscles (SA) were recorded as milivolt.
Range of motion | Through study completion, an average of 6 months
  Ultium Motion (Noraxon) range of motion sensors were utilized to record shoulde rmovements during the PNF D2 shoulder flexion exercise in three different planes of motion via flexion, abduction, and external rotation. "Degree" was used as unit measure to record the range of motion.

SECONDARY OUTCOMES:
Age | Through study completion, an average of 6 months
  Participants filled demographics survey including age in years.
Height | Through study completion, an average of 6 months
  the participants filled demographics survey including height in inches
weight | Through study completion, an average of 6 months
  The participants filled demographics survey including weight in pound
The Borg Rating of Perceived Exertion scale | Through study completion, an average of 6 months
  The Borg Rating of Perceived Exertion scale that ranges from 6 to 20 where 6 means "no exertion at all" and 20 means "maximal exertion." was used to determine the level of physical activity during therapeutic exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Edeer, PT, PhD, Principal Investigator — Dominican University New York
Locations (1):
- Dominican University New York, Doctor of Physical Therapy Program, Orangeburg, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lupinacci G, Gatti G, Melegari C, Fontana S. Interactive design of patient-oriented video-games for rehabilitation: concept and application. Disabil Rehabil Assist Technol. 2018 Apr;13(3):234-244. doi: 10.1080/17483107.2017.1306592. Epub 2017 Apr 11. PMID 28398175
- [Result] Ekblom MM, Eriksson M. Concurrent EMG feedback acutely improves strength and muscle activation. Eur J Appl Physiol. 2012 May;112(5):1899-905. doi: 10.1007/s00421-011-2162-2. Epub 2011 Sep 16. PMID 21922262
- [Result] Morais N, Ferreira J, Gordo J, et al. A diagonal movement pattern of arm elevation and depression in overhead throwing athletes: An exploratory kinematic analysis for Clinical Application. Applied Sciences. 2023 Sept 26;13(19):1-15. doi:10.3390/app131910691
- [Result] Forbush SW, Bandy WD, Garrison MK, Graves LC, Roberts R. TESTING INFRASPINATUS AND DELTOID MUSCLES WITH NEW TECHNIQUE TO DECREASE DELTOID ACTIVITY DURING TESTING USING EMG ANALYSIS. Int J Sports Phys Ther. 2018 Aug;13(5):896-904. PMID 30276022
- [Result] Januario LB, Cid MM, Zanca GG, Mattiello SM, Oliveira AB. Serratus anterior sEMG - sensor placement and test position for normalization purposes during maximal and submaximal exertions. Med Eng Phys. 2022 Mar;101:103765. doi: 10.1016/j.medengphy.2022.103765. Epub 2022 Feb 8. PMID 35232545
- [Result] Huang HY, Lin JJ, Guo YL, Wang WT, Chen YJ. EMG biofeedback effectiveness to alter muscle activity pattern and scapular kinematics in subjects with and without shoulder impingement. J Electromyogr Kinesiol. 2013 Feb;23(1):267-74. doi: 10.1016/j.jelekin.2012.09.007. Epub 2012 Nov 2. PMID 23123099
- [Result] Cheng, L., Li, J., Guo, A. et al. Recent advances in flexible noninvasive electrodes for surface electromyography acquisition. npj Flex Electron 7, 39 (2023). https://doi.org/10.1038/s41528-023-00273-0
- [Result] Szczepan S, Zaton K, Fernandez FC, et al. The effects of concurrent visual versus verbal feedback on swimming strength task execution. Balt J Health Phys Act. 2018;10(4):61-71. doi:10.29359/BJHPA.10.4.05.
- [Result] Chen MJ, Fan X, Moe ST. Criterion-related validity of the Borg ratings of perceived exertion scale in healthy individuals: a meta-analysis. J Sports Sci. 2002 Nov;20(11):873-99. doi: 10.1080/026404102320761787. PMID 12430990
- [Result] Chen C, Weyland S, Fritsch J, Woll A, Niessner C, Burchartz A, Schmidt SCE, Jekauc D. A Short Version of the Physical Activity Enjoyment Scale: Development and Psychometric Properties. Int J Environ Res Public Health. 2021 Oct 20;18(21):11035. doi: 10.3390/ijerph182111035. PMID 34769552
- [Result] Grime A, Daines S, Pringle L, et al. The within-day reliability of scapular and shoulder EMG measurements in asymptomatic individuals during shoulder abduction. NZJP. 2023;46(2):67-72. doi:10.15619/NZJP/46.2.02.
- [Result] Alizadehkhaiyat O, Hawkes DH, Kemp GJ, Frostick SP. ELECTROMYOGRAPHIC ANALYSIS OF SHOULDER GIRDLE MUSCLES DURING COMMON INTERNAL ROTATION EXERCISES. Int J Sports Phys Ther. 2015 Oct;10(5):645-54. PMID 26491615
- [Result] Campanini I, Disselhorst-Klug C, Rymer WZ, Merletti R. Surface EMG in Clinical Assessment and Neurorehabilitation: Barriers Limiting Its Use. Front Neurol. 2020 Sep 2;11:934. doi: 10.3389/fneur.2020.00934. eCollection 2020. PMID 32982942
- [Result] San Juan JG, Gunderson SR, Kane-Ronning K, Suprak DN. Scapular kinematic is altered after electromyography biofeedback training. J Biomech. 2016 Jun 14;49(9):1881-1886. doi: 10.1016/j.jbiomech.2016.04.036. Epub 2016 May 3. PMID 27161990
- [Result] Vitali RV, Barone VJ, Ferris J, Stirling LA, Sienko KH. Effects of Concurrent and Terminal Visual Feedback on Ankle Co-Contraction in Older Adults during Standing Balance. Sensors (Basel). 2021 Nov 2;21(21):7305. doi: 10.3390/s21217305. PMID 34770611
- [Result] Youdas JW, Arend DB, Exstrom JM, Helmus TJ, Rozeboom JD, Hollman JH. Comparison of muscle activation levels during arm abduction in the plane of the scapula vs. proprioceptive neuromuscular facilitation upper extremity patterns. J Strength Cond Res. 2012 Apr;26(4):1058-65. doi: 10.1519/JSC.0b013e31822e597f. PMID 22446675
- [Result] Knippenberg E, Verbrugghe J, Lamers I, Palmaers S, Timmermans A, Spooren A. Markerless motion capture systems as training device in neurological rehabilitation: a systematic review of their use, application, target population and efficacy. J Neuroeng Rehabil. 2017 Jun 24;14(1):61. doi: 10.1186/s12984-017-0270-x. PMID 28646914
- [Result] Lee HL, Khairunizam W, Cahyadi BN, et al. Progress monitoring in upper limb stroke rehabilitation by using muscle activation and hand speed. J Phys: Conf Ser. 2020;1529(4):042019. doi:10.1088/1742-6596/1529/4/042019
- [Result] Fuertes Munoz G, Mollineda RA, Gallardo Casero J, Pla F. A RGBD-Based Interactive System for Gaming-Driven Rehabilitation of Upper Limbs. Sensors (Basel). 2019 Aug 9;19(16):3478. doi: 10.3390/s19163478. PMID 31395817
- [Result] Zaidi S, Ahamad A, Fatima A, Ahmad I, Malhotra D, Al Muslem WH, Abdulaziz S, Nuhmani S. Immediate and Long-Term Effectiveness of Proprioceptive Neuromuscular Facilitation and Static Stretching on Joint Range of Motion, Flexibility, and Electromyographic Activity of Knee Muscles in Older Adults. J Clin Med. 2023 Mar 30;12(7):2610. doi: 10.3390/jcm12072610. PMID 37048693
- [Result] Witt D, Talbott N, Kotowski S. Electromyographic activity of scapular muscles during diagonal patterns using elastic resistance and free weights. Int J Sports Phys Ther. 2011 Dec;6(4):322-32. PMID 22163094